CLINICAL TRIAL: NCT04713423
Title: Oral and Perioral Herpes Simplex Virus Infection Type I in a Five-month-old Infant: A Case Report
Status: Completed | Type: Observational
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Ashwag Yagoub Aloyouny, Senior registrar of Oral Medicine, Princess Nourah Bint Abdulrahman University
Other Study IDs: PrincessNBAU
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Herpes Simplex Virus Infection
Keywords: Herpetic gingivostomatitis; Herpes simplex virus; Perioral lesions; Infants; Case report; Herpes simplex virus type 1; Oral lesions
MeSH Terms: conditions — Herpes Simplex; Stomatitis, Herpetic | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnosis and treatment of the case — The infant was transferred to a hospital for better management of her infection. She was immediately started on intravenous acyclovir (20 mg/kg/6 h/5 d) while acetaminophen suppositories (80 mg/8 h/5 d) were given to lower her body temperature. In addition, other palliative drugs, such as diphenhydramine syrup (12.5 mg/5 mL, 2.5 mL orally) once-a-night for five days, were given to ease the effort of drinking and to aid in achieving good sleep. Upon completion of five days of therapy, the patient showed complete recovery and was subsequently discharged from the hospital free from symptoms.

SUMMARY:
A five-month-old healthy girl who presented with painful herpetic gingivostomatitis and perioral vesicles.

DETAILED DESCRIPTION:
The investigators present the case of a five-month-old healthy girl who presented with painful herpetic gingivostomatitis and perioral vesicles. The investigators discuss the pathophysiology of primary herpes simplex virus infection and the effect of maternal antibodies on the infant's immune system. In addition, the investigators explain the diagnosis, management, and prognosis of herpes simplex virus infection in young infants.

ELIGIBILITY:
Inclusion Criteria:

* Five-months-old infants or younger

Exclusion Criteria:

* Six-months-old infants or older

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a case report study
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Health condition | one week
  Number of tests were performed and different drugs were administered

CONTACTS AND LOCATIONS:
Overall Officials: Ashwag Y Aloyouny, Principal Investigator — Princess Nourah Bint Abdulrahman University
Locations (1):
- Princess Nourah Bint Abdulrahman University, Riyadh, Saudi Arabia